CLINICAL TRIAL: NCT06727474
Title: Evolution of Quality of Life, Functional Capacity, Nutritional Status and Return to Work Activity in Patients Admitted for Severe Pneumonia Due to COVID 19 Requiring Invasive Mechanical Ventilation
Brief Title: Clinical and Funtional Caracteristics of Patients Admitted for Severe Pneumonia Due to COVID 19.
Acronym: EQOL-COVID
Status: Completed | Type: Observational
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Sponsor
Other Study IDs: 01-2024
Record Dates: First submitted 2024-12-02; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Post-intensive Care Syndrome; COVID-19
Keywords: COVID-19; health-related quality of life; functional capacity; nutritional status; reintegration into work; post-intensive care syndrome
MeSH Terms: conditions — postintensive care syndrome; COVID-19 | interventions — Visual Analog Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow up cohort: Discharged alive from the ICU and admitted to the follow-up program. Programed scheduled visits, which included an evaluation at one month, six months, and one year after hospital discharge
  Interventions: Diagnostic Test: Health-Related Quality of Life (HRQoL) with EQ-5D-3L

INTERVENTIONS:
Diagnostic Test: Health-Related Quality of Life (HRQoL) with EQ-5D-3L — The EQ-5D-3L and EQ-VAS questionnaires, administered at all visits, evaluated five dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Responses generated a Health Status sequence and calculated the EQ-5D-3L Index. A visual analogue scale (VAS) rated health from 0 (worst) to 100 (best). Functional capacity was assessed using the Katz Index (IK) and Timed Up and Go (TUG), which measured the time to rise from a chair, walk 3 meters, and return. Anthropometric variables, measured by the same researcher (LP) at 1 month and 1 year, included limb circumferences using specific techniques. Muscle strength, evaluated with the EF-MRC scale, involved verbal commands for movement tests. Calf circumference was measured on the largest circumference area. Living conditions and work reintegration were recorded. Health issues detected during follow-up were referred to the clinic's coordinating physician for appropriate care.
  Other Names: EuroQol-5D VAS (Analog visual scale); Medical Reseacrh Council Strength Scale; Katz index for functional independence; Timed Up to Go test; Waist Circunference; Brachial Circumference; Calf Circumference

SUMMARY:
This research protocol aims to evaluate the impact of severe COVID-19 pneumonia requiring invasive mechanical ventilation (IMV) on health-related quality of life (HRQoL), functional capacity, muscle strength, and nutritional status one year after discharge from the ICU. The study is analytical, longitudinal, and prospective, involving patients over 18 years who received IMV for more than 72 hours and were discharged alive. Primary outcomes include changes in HRQoL (assessed using EQ-5D-3L and VAS), functional capacity (Katz Index and Timed Up and Go test), muscle strength (MRC scale), and nutritional status (BMI and limb circumferences). Secondary outcomes include time to return to work and one-year mortality. Data collection occurs at discharge and at one, six, and twelve months post-discharge. Statistical analyses involve descriptive statistics and longitudinal comparisons using Friedman and Dunn-Bonferroni tests. Ethical approval has been secured, and patient anonymity will be ensured. The protocol emphasizes multidisciplinary follow-up to identify and address physical and psychological sequelae effectively.

DETAILED DESCRIPTION:
This study aims to evaluate the long-term impact of severe COVID-19 pneumonia on patients requiring invasive mechanical ventilation (IMV) for more than 72 hours. Specifically, it examines health-related quality of life (HRQoL), functional capacity, muscle strength, nutritional status, and work reintegration at various time points up to one year after ICU discharge. Additionally, it assesses one-year post-hospital discharge mortality and the time required for patients to return to work.

The study employs a prospective, longitudinal design, following a cohort of patients aged 18 years and older discharged alive from the ICU. Participants were selected based on strict inclusion criteria, such as confirmed COVID-19 pneumonia requiring IMV for over 72 hours and the ability to provide informed consent. Exclusion criteria included cognitive impairment, prior tracheostomy, or pre-existing indications for home mechanical ventilation. The population was evaluated across four defined time points: before hospital discharge (Visit 0), at one month (Visit 1), at six months (Visit 2), and at one year post-discharge (Visit 3).

Clinical, demographic, and functional data were collected through validated tools. HRQoL was assessed using the EQ-5D-3L index and visual analog scale (VAS), while functional capacity was measured with the Katz Index and the Timed Up and Go (TUG) test. Muscle strength was evaluated using the Medical Research Council (MRC) scale, and nutritional status was determined through BMI and anthropometric measurements, including arm, waist, and calf circumferences. Additional data included work reintegration and mortality outcomes, tracked through patient interviews and medical records.

Data analysis employed robust statistical methods to identify trends and differences across time points. Descriptive statistics summarized demographic and baseline clinical characteristics. Longitudinal comparisons were conducted using repeated measures ANOVA or Friedman tests, with post-hoc analysis (Bonferroni or Dunn-Bonferroni) to evaluate significant pairwise differences. For comparisons involving only two time points, paired t-tests or Wilcoxon signed-rank tests were used as appropriate. All analyses adhered to a significance threshold of p < 0.05, and data visualization was performed using SPSS and R software packages.

Ethical considerations were rigorously maintained. The study was approved by the Ethics Committee of the Hospital Nacional Prof. Alejandro Posadas, and informed consent was obtained from all participants. Patient anonymity was preserved using unique coded identifiers, and all procedures complied with established guidelines for research integrity and participant safety.

Preliminary results indicate significant improvements in HRQoL, functional capacity, and muscle strength over the one-year follow-up period. However, persistent challenges such as delayed work reintegration and moderate mortality rates highlight the complex recovery trajectory of critically ill COVID-19 survivors. This study underscores the importance of structured, multidisciplinary follow-up programs to address the physical, nutritional, and psychosocial needs of this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* discharged alive from the ICU
* over 18 years of age
* diagnosis of admission or reason for hospitalization in the ICU of pneumonia due to COVID-19, all had to have confirmed the presence of SARS-CoV-2 as a causative agent by a positive result of a real-time reverse transcriptase polymerase chain reaction assay with nasopharyngeal swab samples or tracheal aspirated respiratory airway sample.
* have received invasive mechanical ventilatory assistance for more than 72 hours
* the patient or a close family member had agreed to participate in the study by signing the informed consent.

Exclusion Criteria:

* patients in jail at the time of admission to the ICU.
* history of dementia or cognitive impairment.
* those who already had a previous tracheostomy for any reason
* prior to admission to the ICU indication of prolonged mechanical ventilation at home or in a chronic care institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the period between June and December 2020, all patients who were discharged alive from the ICU, were referred to the general hospitalization ward and were discharged from hospital were included
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | 1 year
  The percentage of change in health-related quality of life (HRQoL) will be measured. This is a multidimensional concept that assesses the physical, psychological and social aspects of an individual's well-being, specifically as it is influenced by their health status.
  This study assesses health-related quality of life using the EuroQol-5 Dimension 3 Level (EQ-5D-3L) questionnaire. The EQ-5D-3L includes a descriptive system that covers five domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analogue scale (VAS) that ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
  Unit of measurement: EQ-5D-3L Index: a calculated score derived from the descriptive system that reflects overall health-related quality of life.
  EQ-5D VAS: a self-reported numerical score that represents perceived health status.
Functional capacity | 1 year
  Measured through The Katz Index assesses functional independence in six basic activities of daily living: bathing, dressing, toileting, transferring, continence, and feeding.
  Unit of Measure: Score on the Katz Index (range 0-6, where 6 indicates full independence).
  Outcome Measure 2: Functional Mobility - Timed Up and Go (TUG) Test The TUG test measures functional mobility by recording the time (in seconds) it takes for a participant to stand from a seated position, walk 3 meters, turn around, walk back, and sit down.
  Unit of Measure:
  Time in seconds.
  Time Frame:
  Assessed at three time points: at one month, at six months, and one year post-discharge (not applicable before hospital discharge as participants may not be ambulatory).
Functional capacity | 1 year
  Measured through Time up to go (TUG) test. The TUG test measures functional mobility by recording the time (in seconds) it takes for a participant to stand from a seated position, walk 3 meters, turn around, walk back, and sit down.
  Unit of Measure: Time in seconds. The Katz Index assesses functional independence in six basic activities of daily living: bathing, dressing, toileting, transferring, continence, and feeding.
  Unit of Measure: Score on the Katz Index (range 0-6, where 6 indicates full independence).
Muscle Strength | 1 year
  Measured through Medical Research Council (MRC) Strength Scale: The MRC Strength Scale evaluates muscle strength across six muscle groups in both upper and lower limbs. Each group is scored on a 6-point scale ranging from 0 (no movement) to 5 (normal strength), with a total score ranging from 0 to 60.
  Unit of Measure:
  Total score on the MRC Strength Scale (range 0-60, where higher scores indicate better muscle strength).
Anthropometric variables - Body mass index | 1 year
  current Weight in kilograms (kg) and Height in meters (m) for calculation of body mass index (BMI). BMI is calculated as weight (kg) divided by height squared (m²).
  Unit of Measure: BMI in kg/m².
Anthropometric variables - | 1 year
  WC is measured using a non-stretchable measuring tape at the midpoint between the last rib and the iliac crest.
  Unit of Measure: Circumference in centimeters (cm).
Anthropometric variables - Arm Circumference (AC) | 1 year
  AC is measured at the midpoint between the acromion and the olecranon. Unit of Measure: Circumference in centimeters (cm).
Anthropometric variables - Calf Circumference (CC) | 1 year
  CC is measured at the point of maximum circumference of the calf. Unit of Measure: Circumference in centimeters (cm).

SECONDARY OUTCOMES:
Number of patients who returned to work | 1 year
  patients who had stated that they had been working prior to hospitalization were asked about the return to work.
  Unit of Measure: Number of participants (count).
Number of Participants Who Died During the One-Year Follow-Up | 1 year
  Mortality was determined by reviewing medical records and contacting patients or their families if they missed a scheduled clinic visit. The reason for non-attendance was investigated, and deaths were recorded when confirmed.
  Unit of Measure: Number of participants (count).

CONTACTS AND LOCATIONS:
Locations (1):
- Ladislao Diaz Ballve, Haedo, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 1 year after finalization
Access Criteria: contact principal investigator via e-mail

REFERENCES:
- [Result] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Result] Demoule A, Morawiec E, Decavele M, Ohayon R, Malrin R, Galarza-Jimenez MA, Laveneziana P, Morelot-Panzini C, Similowski T, De Rycke Y, Gonzalez-Bermejo J. Health-related quality of life of COVID-19 two and 12 months after intensive care unit admission. Ann Intensive Care. 2022 Feb 20;12(1):16. doi: 10.1186/s13613-022-00991-0. PMID 35184214
- [Result] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Result] Wang X, Xu H, Jiang H, Wang L, Lu C, Wei X, Liu J, Xu S. Clinical features and outcomes of discharged coronavirus disease 2019 patients: a prospective cohort study. QJM. 2020 Sep 1;113(9):657-665. doi: 10.1093/qjmed/hcaa178. PMID 32442308
- [Result] Pironi L, Sasdelli AS, Ravaioli F, Baracco B, Battaiola C, Bocedi G, Brodosi L, Leoni L, Mari GA, Musio A. Malnutrition and nutritional therapy in patients with SARS-CoV-2 disease. Clin Nutr. 2021 Mar;40(3):1330-1337. doi: 10.1016/j.clnu.2020.08.021. Epub 2020 Aug 27. PMID 32900518
- [Result] Whittle J, Molinger J, MacLeod D, Haines K, Wischmeyer PE; LEEP-COVID Study Group. Persistent hypermetabolism and longitudinal energy expenditure in critically ill patients with COVID-19. Crit Care. 2020 Sep 28;24(1):581. doi: 10.1186/s13054-020-03286-7. No abstract available. PMID 32988390
- [Result] Alvarez-Hernandez J, Matia-Martin P, Cancer-Minchot E, Cuerda C; NUTRICOVID study group of SENDIMAD. Long-term outcomes in critically ill patients who survived COVID-19: The NUTRICOVID observational cohort study. Clin Nutr. 2023 Oct;42(10):2029-2035. doi: 10.1016/j.clnu.2023.08.008. Epub 2023 Aug 16. PMID 37659250
- [Result] Kamdar BB, Suri R, Suchyta MR, Digrande KF, Sherwood KD, Colantuoni E, Dinglas VD, Needham DM, Hopkins RO. Return to work after critical illness: a systematic review and meta-analysis. Thorax. 2020 Jan;75(1):17-27. doi: 10.1136/thoraxjnl-2019-213803. Epub 2019 Nov 8. PMID 31704795
- [Result] Das Neves AV, Vasquez DN, Loudet CI, Intile D, Saenz MG, Marchena C, Gonzalez AL, Moreira J, Reina R, Estenssoro E. Symptom burden and health-related quality of life among intensive care unit survivors in Argentina: A prospective cohort study. J Crit Care. 2015 Oct;30(5):1049-54. doi: 10.1016/j.jcrc.2015.05.021. Epub 2015 Jun 3. PMID 26105747